CLINICAL TRIAL: NCT01375023
Title: Allogenic Haematopoietic Cell Transplantation Using a Non-myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin for Patients With Refractory "Triple Negative" Breast Cancer
Brief Title: Allogenic Haematopoietic Cell Transplantation for Patients With Refractory "Triple Negative" Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very low accrual rate
Sponsor: European Institute of Oncology (Other)
Collaborators: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO S438/508; 2008-006262-28 (EudraCT Number)
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: Allogenic Haematopoietic Cell Transplantation; Total Lymphoid Irradiation; Anti-Thymocyte Globulin; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Radiotherapy; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-Thymocyte Globulin+radiotherapy (Experimental): triple negative breast cancer patients treated with radiation and Anti-Thymocyte Globulin iv
  Interventions: Radiation: Radiotherapy; Biological: Anti-Thymocyte Globulin

INTERVENTIONS:
Radiation: Radiotherapy — daily radiation therapy for 10 days, total dose of 80 cGY
Biological: Anti-Thymocyte Globulin — 1.5 mg/kg/day, IV from day -11 through day -7 before transplantation
  Other Names: Thymoglobuline

SUMMARY:
The purpose of this study is to evaluate the engraftment, toxicity and anti-tumour activity of allogeneic peripheral blood progenitor cell (PBPC) transplantation using TLI/ATG conditioning regimen in patients with refractory "Triple Negative" breast cancer.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer among women and approximately 45% of breast cancer patients develop metastatic disease that generally remains incurable with a median survival of approximately 18 to 24 months. A subpopulation emerging as having particularly poor prognosis is patients who have disease that is receptor negative for oestrogen, progestin and HER2/neu (triple receptor negative). Since no effective therapy is available in this setting of patients, the investigators propose allogeneic haematopoietic cell transplantation.

Recent advances in allogeneic haematopoietic cell transplantation (HCT) have led to reduced intensity preparative regimens that are non-myeloablative and permit the development of sustained donor chimerism. As a result, regimen related organ toxicities (RROT), and consequently non-relapse mortality has been reduced. However, the incidence of acute and chronic graft-versus-host disease (aGVHD and cGVHD, respectively) has remained a major complication. Pre-clinical data, developed by the Stanford group, established that nonmyeloablative conditioning with total lymphoid irradiation (TLI) combined with depletive anti-T cell antibodies protects against GVHD by skewing peripheral T cell subsets to favour suppressive regulatory T cells. The current proposal is a Phase II study evaluating safety and activity of the allogeneic peripheral blood progenitor cell (PBPC) transplantation using TLI/ATG conditioning regimen, the kinetics of donor haematopoietic cell engraftment and chimerism, the incidence and severity of acute GVHD following allogeneic transplantation using the novel preparative regimen of TLI combined with antithymocyte globulin (ATG). Patients with triple negative breast cancer will be considered for transplantation using donor grafts from HLA-matched related donors. The preparative regimen of TLI combined with ATG is expected to result in high levels of sustained donor haematopoietic cell engraftment with a significantly reduced incidence of acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer with evidence of unresectable, locally recurrent, or metastatic disease. Locally recurrent disease must not be amenable to resection or radiation therapy with curative intent.
* Documentation of estrogen and progestin receptor (ER/PR) negative status and HER2/neu receptor negative status (ie, FISH or CISH (where approved) negative or immunohistochemistry 0 or +1).
* Prior treatment with an anthracycline, a taxane and alkylating agents alone or in combination in the neoadjuvant, adjuvant or metastatic disease setting.
* Prior treatment with chemotherapy as follows: Receipt of adjuvant chemotherapy with RECIST (appendix B) defined disease progression documented during treatment or disease relapse within 6 months of last treatment, OR Receipt of chemotherapy in the first-line advanced disease setting with RECIST defined disease stable or progression documented during treatment, or, if the patient completed treatment with objective disease response, documented disease progression after discontinuing treatment. Patients entering the study on the basis of this criterion may have also previously received neo adjuvant or adjuvant treatment with chemotherapy.
* Measurable disease as per RECIST. Measurable lesions that have been previously radiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.
* Male or female.
* Patients age > 18 and < 70 years.
* ECOG performance status 0-2.
* Resolution of all acute toxic effects of prior therapy or surgical procedures to grade ≤1 (except alopecia).
* Life expectancy >6 months.
* A fully HLA-identical sibling donor is available. Patients with one antigen mismatched donors can be considered but only after discussion with the transplant team and the Principal Investigator.
* The definitions of minimum adequacy for organ function required prior to study entry are as follows: serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy; total serum bilirubin ≤1.5 x ULN; serum albumin ≥3.0 g/dL; absolute neutrophil count (ANC) ≥1500/μL; platelets ≥100,000/μL; haemoglobin ≥9.0 g/dL; serum creatinine ≤1.5 x ULN
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Uncontrolled CNS involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Organ dysfunction defined as follows: cardiac ejection fraction <30% or uncontrolled cardiac failure; pulmonary: DLCO <40% predicted; liver: elevation of bilirubin to > 1.5 X ULN and/or transaminases >5x the upper limit of normal Renal: Serum creatinine >1.5 x ULN
* ECOG performance status > 2
* Patients with poorly controlled hypertension on multiple antihypertensives
* Documented fungal disease that is progressive despite treatment
* Viral infections: HIV positive patients. Hepatitis B and C positive patients will be evaluated on a case by case basis
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Any previous or current malignancy at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix and adequately treated basal or squamous cell carcinoma of the skin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response to treatment according to RECIST criteria | 90 after the baseline
  Response to treatment according to RECIST criteria evaluated after 90 days from baseline

SECONDARY OUTCOMES:
graft versus host disease (GVHD) | Time Frame: Day +365
  incidence and severity of GVHD after one year from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Pastano, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Background] Storb RF, Champlin R, Riddell SR, Murata M, Bryant S, Warren EH. Non-myeloablative transplants for malignant disease. Hematology Am Soc Hematol Educ Program. 2001:375-91. doi: 10.1182/asheducation-2001.1.375. PMID 11722994
- [Background] Ueno NT, Rondon G, Mirza NQ, Geisler DK, Anderlini P, Giralt SA, Andersson BS, Claxton DF, Gajewski JL, Khouri IF, Korbling M, Mehra RC, Przepiorka D, Rahman Z, Samuels BI, van Besien K, Hortobagyi GN, Champlin RE. Allogeneic peripheral-blood progenitor-cell transplantation for poor-risk patients with metastatic breast cancer. J Clin Oncol. 1998 Mar;16(3):986-93. doi: 10.1200/JCO.1998.16.3.986. PMID 9508181
- [Background] Sandmaier BM, Mackinnon S, Childs RW. Reduced intensity conditioning for allogeneic hematopoietic cell transplantation: current perspectives. Biol Blood Marrow Transplant. 2007 Jan;13(1 Suppl 1):87-97. doi: 10.1016/j.bbmt.2006.10.015. PMID 17222778